CLINICAL TRIAL: NCT04760691
Title: A Phase I Trial for the Evaluation of the Two-way Pharmacokinetic-pharmacodynamic (PD) Interaction of Gender Affirming Exogenous Estrogen (With Testosterone Suppression) on TDF/FTC PrEP in Transgender Women (TGW)
Brief Title: Pre-Exposure Prophylaxis (PrEP)- Gender Affirming Hormone Therapy (GAHT) Interactions in TGW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00203162; R01AI145675 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Prophylaxis; Transgender
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; Leuprolide; Estradiol; Estrogens; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pre-Exposure Prophylaxis (PrEP) only (Active Comparator): Truvada one tablet by mouth daily
  Interventions: Drug: Truvada alone
- PrEP plus Gonadotropin Releasing Hormone (GnRH) Agonist (Experimental): Truvada one tablet by mouth daily Leuprolide 11.25 milligrams (mg) intramuscular (im) injection once
  Interventions: Drug: Truvada plus Leuprolide
- PrEP plus Low Dose Estrogen (Experimental): Truvada one tablet by mouth daily Estradiol 1 milligram by mouth daily x 2 weeks
  Interventions: Drug: Truvada plus Estradiol 1 mg
- PrEP plus High Dose Estrogen (Experimental): Truvada one tablet by mouth daily Estradiol 6 milligrams (mg) by mouth daily x 2 weeks
  Interventions: Drug: Truvada plus Estradiol 6 mg
- High Dose Estrogen (Experimental): Estradiol 6 mg by mouth daily x 2 weeks
  Interventions: Drug: Estradiol 6 mg alone

INTERVENTIONS:
Drug: Truvada alone — TDF/FTC 300 mg (milligrams) / 200 mg by mouth once daily
  Other Names: tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)
  Arms: Pre-Exposure Prophylaxis (PrEP) only
Drug: Truvada plus Leuprolide — TDF/FTC 300mg/ 200 mg by mouth once daily Leuprolide 11.25 mg im once
  Other Names: Truvada plus Lupron
  Arms: PrEP plus Gonadotropin Releasing Hormone (GnRH) Agonist
Drug: Truvada plus Estradiol 1 mg — TDF/FTC 300mg/ 200 mg by mouth once daily Estradiol 1 mg by mouth once daily
  Other Names: Truvada plus low dose estrogen
  Arms: PrEP plus Low Dose Estrogen
Drug: Truvada plus Estradiol 6 mg — TDF/FTC 300mg/ 200 mg by mouth once daily Estradiol 3 mg by mouth twie daily
  Other Names: Truvada plus high dose estrogen
  Arms: PrEP plus High Dose Estrogen
Drug: Estradiol 6 mg alone — Estradiol 3 mg by mouth twice daily
  Other Names: Estradiol 6 mg
  Arms: High Dose Estrogen

SUMMARY:
This is a research study to determine the best way to dose Truvada®, an oral medication licensed to be taken as Pre-Exposure Prophylaxis (PrEP) to prevent HIV infection, in transgender women who are also taking feminizing hormones. The duration of the study is about 4 months, and involves a screening visit, a baseline visit with colon biopsies and kidney function testing, and several outpatient visits, including 5 intensive sampling visits that last about 9 hours and involve colon biopsies, kidney function testing and other blood specimen collections.

After the baseline visit, participants will start on PrEP, daily Truvada® pills, and will continue on the Truvada® for 5 weeks. Participants will then receive either an injection of Lupron, oral low-dose estradiol or oral high-dose estradiol, which will be taken along with the Truvada® PrEP for 1-2 weeks before returning for an intensive sampling visit.

DETAILED DESCRIPTION:
The PrEP-GAHT Interactions in TGW protocol is a phase 1, open label study to compare the safety, PK and PD of five sequential phases of PrEP administration in the presence or absence of testosterone-reducing therapies or dose-escalated estrogen therapy. Each participant will undergo a Screening Visit to evaluate eligibility.

Following Baseline evaluation, eligible participants will receive 300 milligrams (mg) TDF/200 mg FTC (Truvada®) once daily for seven days, using direct observation approaches, to achieve steady state drug PrEP concentrations. After one week of therapy, participants will undergo intensive PK analysis as well as collection of colorectal biopsies for PD testing (PK1). During the PK-intensive day, iohexol will be administered intravenously for the empirical determination of renal function and measured glomerular filtration rate (mGFR). While concurrently on PrEP, participants will then be intramuscularly administered depot leuprolide acetate (11.25 mg Lupron®). Two weeks post-injection, when testosterone concentrations are far below the lower limit of normal of total testosterone in men (typically < 200 ng/dL, or < 2 ng/mL), sampling for PK, PD, and renal function will be performed (PK2).

Participants will then immediately begin low-dose oral estrogen therapy (1 mg 17β-estradiol) in conjunction with PrEP for one week, at which time samples will be collected for the analyses described above (PK3). While still on PrEP, participants will then transition to high-dose estrogen therapy (6 mg 17β-estradiol) for the remainder of the study. One week post-high dose estrogen therapy in the presence of PrEP, pharmacologic and renal samples will be collected for analysis (PK4). PrEP will then be discontinued, and two weeks later, samples will be collected to assess renal function and hormonal concentrations, and evaluate the presence of any remaining PrEP in plasma, Peripheral Blood Mononuclear Cells (PBMC), or colorectal tissue (though it should be near undetectable levels for most analytes according to the investigators' prior data)(PK5).

Safety assessments, including history/physical, chemistry/hematology labs at screening and interim history will be performed at each study-intensive visit. Additionally, periodic assessments of gender dysphoria will be conducted at baseline and a convenient time during PK visits throughout the study. To ensure compliance, participants will undergo direct observation of dosing each day of the week prior to PK visits, using the aforementioned strategies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Self-identifying as a transgender woman
3. Not currently taking any gender affirming hormonal therapy (GAHT) with a total testosterone concentration of ≥ 200 ng/dL, or willing to abstain from feminizing therapies (including estradiol, spironolactone, progesterone, etc.) until total total testosterone concentrations are ≥ 200 ng/dL. Note: Testosterone may be retested every 2-4 weeks during screening to determine eligibility up to 6 weeks.
4. HIV-1 uninfected at screening as documented by Combo Ag/Ab HIV-1/HIV-2 immunoassay
5. Understand and agree to local STI reporting requirements
6. Able and willing to communicate in English
7. Able and willing to provide written informed consent to take part in the study
8. Able and willing to provide adequate information for locator purposes
9. Able and willing to participate in a directly observed study, which may occur in person, using live streaming or a time stamped video?
10. Availability to return for all study visits, barring unforeseen circumstances
11. Willing to abstain from insertion of anything (drug, enema, penis, or sex toy) in rectum for 72 hours before and 72 hours after each flexible sigmoidoscopy
12. Willing to refrain from aspirin and NSAID use for one week before and after each study biopsy visit
13. Willing and able to use condoms for all Receptive Anal Intercourse (RAI) for the duration of participation
14. Willing and able to participate in a directly observed study, which may occur in person, using live streaming or a time stamped video
15. Has an identified healthcare provider for transgender health management
16. Agree not to participate in other research studies involving drugs and/or medical devices for the duration of the study

Exclusion Criteria:

1. Not currently on any PrEP regimen (e.g., Truvada®, tenofovir alafenamide/ emtricitabine)
2. History of chronic Hepatitis B infection, as documented by positive HBsAg at screening
3. ≥ Grade 2 laboratory abnormality at baseline as defined by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 - July 2017, and Addendum 3 (Rectal Grading Tables for Use in Microbicide Studies)
4. Significant colorectal symptom(s) as determined by medical history or by participant self- report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
5. At screening or within the past 2 months: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal infection requiring treatment per current Centers for Disease Control (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active herpes simplex virus (HSV) lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion. (Note: if an Sexually Transmitted Infection (STI) apart from HIV is detected, the participant will be referred for treatment and can be retested in 30 days and rescreened once.)
6. History of an underlying clinically significant cardiac arrhythmia or renal disease (including creatinine clearance < 60 mL/min using Cockcroft-Gault equation)
7. Serum phosphate < 2.3 mg/dL
8. History of severe or recent cardiac or pulmonary event
9. History of significant gastrointestinal bleeding
10. Current use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], Non-steroidal anti-inflammatory drug [NSAIDs], or Pradaxa®)
11. Use of systemic or anorectal immunomodulatory medications within 4 weeks of enrollment or planned use at any time during study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender women (biologic sex identified male at birth; identifying as female)
Enrollment: 13 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in Tenofovir plasma concentration | Days 7-8, Days 21-22, Days 28-29, Days 35-36, Days 49-50
  Change in Tenofovir plasma concentration measured in nanograms (ng) per milliliter (mL)
Change in Tenofovir-Diphosphate PBMC concentration | Days 7-8, Days 21-22, Days 28-29, Days 35-36, Days 49-50
  Change in tenofovir-diphosphate (TFV-DP) PBMC concentration reported in femtomoles per million cells (fmol/million)
Change in TFV-DP colon tissue concentration | Days 7-8, Days 21-22, Days 28-29, Days 35-36, Days 49-50
  Change in TFV-DP colon tissue concentration reported in fmol/million

SECONDARY OUTCOMES:
Change in serum estradiol concentration | Days 7, 21, 28, 35, 49
  Change in serum estradiol reported in picograms (pg) per mL
Change in serum free testosterone concentration | Days 7, 21, 28, 35, 49
  Serum free testosterone reported in nanograms per deciliter (ng/dL)
Change in serum total testosterone concentration | Days 7, 21, 28, 35, 49
  Change in serum total testosterone reported in ng/dL
Change in Serum luteinizing hormone (LH) concentration | Days 7, 21, 28, 35, 49
  Change in serum LH reported in milli-international units per milliliter (mIU/mL)
Change in serum follicular stimulating hormone (FSH) | Days 7, 21, 28, 35, 49
  Change in serum FSH reported in mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Marzinke, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine Drug Development Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No